CLINICAL TRIAL: NCT04157335
Title: A Multicentre, Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Phase 3 Efficacy and Safety Study of Benralizumab in Patients With Eosinophilic Chronic Rhinosinusitis With Nasal Polyps (ORCHID)
Brief Title: Efficacy and Safety Study of Benralizumab in Patient With Eosinophilic Chronic Rhinosinusitis With Nasal Polyps (ORCHID)
Acronym: ORCHID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has a double-blind period and an open-label period. The study did not meet its primary endpoints after the primary LSLV and the decision was taken to terminate the study early.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3252C00002; 2023-507987-38-00 (Registry Identifier: CTIS); 2021-000267-72 (EudraCT Number)
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Nasal Polyposis; Eosinophilic Chronic Rhinosinusitis
Keywords: Benralizumab; Eosinophilic Chronic Rhinosinusitis with Nasal Polyps; Nasal Polyps; Asthma
MeSH Terms: conditions — Nasal Polyps; Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab administered subcutaneously
  Interventions: Biological: Benralizumab 30 mg
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Biological: Matched placebo

INTERVENTIONS:
Biological: Benralizumab 30 mg — Benralizumab is 30 mg/ml solution for injection in accessorized pre-filled syringe, 1 ml fill volume.
  Benralizumab 30 mg subcutaneously will be injected every 4 weeks for the first 3 doses (Weeks 0, 4 and 8) and every 8 weeks thereafter (Weeks 16, 24, 32, 40 and 48).
  For OLE, Benralizumab 30 mg subcutaneously will be injected every 4 weeks for the first 3 doses and every 8 weeks for the rest 5 doses. For the patients on Benralizumab treatment during double blind period, placebo will be dosed at the second dose during OLE.
  Arms: Benralizumab
Biological: Matched placebo — Matching placebo solution for injection in accessorized pre-filled syringe. 1 ml fill volume.
  Matching placebo subcutaneously will be injected every 4 weeks for the first 3 doses (Weeks 0, 4 and 8) and every 8 weeks thereafter (Weeks 16, 24, 32, 40 and 48).
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, international, multicenter, Phase 3 study to evaluate the efficacy and safety of repeat dosing of benralizumab 30 mg administered subcutaneously (SC) versus placebo in patients with severe nasal polyposis.

DETAILED DESCRIPTION:
Approximately 250 patients will be randomized to receive benralizumab 30 mg SC or matching placebo. After enrolment, eligible patients will enter a 6-week screening/run in period. Patients who meet eligibility criteria will be randomised 1:1 at Week 0 (Day 0) to receive either placebo or benralizumab 30 mg SC every 4 weeks for the first 3 doses (Weeks 0, 4 and 8) and every 8 weeks thereafter (Weeks 16, 24, 32, 40 and 48). An end of treatment visit will be conducted at Week 56.All patients who complete the 56-week DB treatment period on investigational product (IP) may be eligible to continue into around one year OLE (Open Label Extension), during which all patients will receive 8 doses of benralizumab 30 mg. Patients in Benra arm during DB period will receive one dummy dose for the second dose during OLE (Open Label Extension). The last study visit will occur at 8 weeks after the last dose of IP (Week 112/FU). Patients who do not enter OLE (Open Label Extension), will have their last study visit at Week 56 (EoDB) for follow-up and without administration of IP.

ELIGIBILITY:
Inclusion criteria:

1. Female or male patients aged 18 to 75 years inclusive
2. Stable Intranasal corticosteroids (INCS) use for at least 4 weeks prior to enrolment and throughout screening and DB period
3. History of treatment with systemic corticosteroids (SCS) or prior surgery for CRSwNP
4. Bilateral sinonasal polyposis with a nasal polyp score (NPS) of 5 at enrolment and randomization (unilateral score of at least 2 for each nostril)
5. Ongoing symptoms for at least 12 weeks prior to enrolment
6. Patient-reported moderate to severe nasal blockage score (NBS) ≥2 at enrolment
7. Bi-weekly mean NBS ≥ 1.5 at randomization
8. SNOT-22 total score ≥ 20 at enrolment and randomization
9. Documented physician-diagnosed asthma
10. Blood eosinophil count of >2% or ≥150/μL at enrolment
11. LMS E≥M for Asian

Exclusion criteria:

1. Any nasal and/or sinus surgery within 3 months prior to enrolment
2. Patients with conditions that makes them non evaluable for the co-primary efficacy endpoint including but not limited to:

   * Unilateral antrochoanal polyps
   * Nasal septal deviation that occludes at least one nostril
   * Current rhinitis medicamentosa
   * Allergic fungal rhinosinusitis or allergic fungal sinusitis;
3. Clinically important comorbidities (other eosinophil-driven diseases but CRSwNP) that may put the patient at risk, or may confound interpretation of clinical efficacy and/or safety results
4. Receipt of SCS for within 4 weeks prior to screening, or a scheduled SCS treatment during the study period.
5. Receipt of any marketed or investigational biologic product within 6 months of enrolment
6. Currently pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Nasal Polyp Burden | Baseline to Week 56
  Change from baseline in endoscopic total nasal polyp score (NPS).
Patient-reported Nasal Blockage (NB) | Baseline to week 56
  Change from baseline in mean nasal blockage score (NBS).

SECONDARY OUTCOMES:
Sense of Smell | Baseline to Week 56
  Change from baseline in difficulty with sense of smell (DSS) score
Sinus Opacification by CT Scan | Baseline to Week 56
  Change from baseline in Lund Mackay score
Disease specific health-related quality of life (HRQoL) | Baseline to Week 56
  Change from baseline in SinoNasal Outcome Test (SNOT-22) score.
Nasal Polyp Surgery | Baseline to Week 56
  Time to first nasal polyp surgery
Systemic corticosteroid (SCS) use | Baseline to Week 56
  Time to first SCS course for CRSwNP
Symptoms associated with CRSwNP | Baseline to Week 56
  Change from baseline in nasal symptom score(s)
Nasal polyp surgery and/or systemic corticosteroids (SCS）for relief of nasal symptoms | Baseline to Week 56
  Time to first NP surgery and/or SCS use for CRSwNP
Nasal polyp surgery and/or systemic corticosteroids (SCS）for relief of nasal symptoms | Baseline to Week 56
  Proportion of patients with NP urgery and/orSCS use for CRSwNP
Nasal polyp surgery | Baseline to Week 56
  Proportion of patients with surgery for CRSwNP
Systemic corticosteroids (SCS) use for relief of nasal symptoms | Baseline to Week 56
  Proportion of patients with SCS use for CRSwNP

OTHER OUTCOMES:
Assessment the safety and tolerability of benralizumab | Baseline to Week 56
  The number of Adverse events (AEs)/serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Prof. Dr., Principal Investigator — Beijing Tongren Hospital
Locations (96):
- United States (15):
  - Research Site, Huntington Beach, California
  - Research Site, Grand Junction, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, White Marsh, Maryland
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Fort Worth, Texas
  - Research Site, McKinney, Texas
  - Research Site, St. George, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aire
  - Research Site, San Fernando
- Australia (3):
  - Research Site, Herston
  - Research Site, Melbourne
  - Research Site, Spearwood
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Chile (3):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
- China (19):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yantai
- France (2):
  - Research Site, Marseille
  - Research Site, Toulouse
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Siófok
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
- Italy (3):
  - Research Site, Catanzaro
  - Research Site, Pisa
  - Research Site, Roma
- Japan (14):
  - Research Site, Chiba
  - Research Site, Fujisawa-shi
  - Research Site, Hiroshima
  - Research Site, Ichikawa-shi
  - Research Site, Iida-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kumamoto
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Moriguchi-shi
  - Research Site, Nagaoka-shi
  - Research Site, Osaka
  - Research Site, Shinjuku-ku
  - Research Site, Yoshida-gun
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Nadarzyn
  - Research Site, Poznan
  - Research Site, Wroclaw
  - Research Site, Łodź
- Russia (3):
  - Research Site, Izhevsk
  - Research Site, Penza
  - Research Site, Saint Petersburg
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Phitsanulok
- Turkey (Türkiye) (4):
  - Research Site, Aydin
  - Research Site, Bakırköy
  - Research Site, Izmir
  - Research Site, Malatya
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614